CLINICAL TRIAL: NCT02360293
Title: Stay Strong: A Physical Activity Program for Afghanistan and Iraq Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRE 12-305
Record Dates: First submitted 2015-01-14; First posted 2015-02-10 (Estimated); Results first posted 2020-01-06 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2019-12

CONDITIONS: Exercise
Keywords: Exercise; App-mediated; Veterans
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stay Strong w/coaching (Experimental): participants in the Stay Strong w/coaching (Experimental) arm are provided a wearable device, scale, telephone coaching, tailored push notifications, personalized goals, and enhanced online/app support.
  Interventions: Behavioral: Stay Strong w/coaching
- Stay Strong (Active Comparator): participants in the Stay Strong (active comparison) arm will only be provided a wearable device with standard online/app support.
  Interventions: Behavioral: Stay Strong

INTERVENTIONS:
Behavioral: Stay Strong w/coaching — Pts randomly placed in the Stay Strong w/coaching group receive an app-mediated physical activity intervention. Pts are asked to wear a physical activity monitoring device and weigh regularly using a Bluetooth scale while participating in the study. Pts will be asked to upload the device data at least weekly and will receive tailored push notifications. Each week the pt will receive a new automatically calculated personalized physical activity goal. Stay Strong coaches will call pts up to 3 times in the first 6-8 weeks of the study to help pts meet physical activity goals including problem solving support. Pts will also be reminded to follow-up with their healthcare provider as needed for the remainder of the 12-month program.
  Arms: Stay Strong w/coaching
Behavioral: Stay Strong — Pts randomly placed in the Stay Strong arm are asked to wear a physical activity monitoring device and weigh regularly using a Bluetooth scale while participating in the study. Pts will be asked to upload the device data at least weekly. Pts will have access to a standard app-mediated intervention that is linked to the wearable device.
  Arms: Stay Strong

SUMMARY:
This project is Project three of a four project Prevention Coaching Lab CREATE grant entitled "Transforming Prevention into Action" aimed at effectively engaging patients and their families to improve their health and medical care.

This project will test the feasibility and effectiveness of the prevention focused, internet mediated healthy lifestyle Stay Strong program tailored to the needs, preferences and demographics of OEF/OIF/OND Veterans.

DETAILED DESCRIPTION:
Veterans from Afghanistan and Iraq (OEF/OIF/OND) are at high risk for becoming overweight and obese. However, existing VA programs are not designed for younger Veterans who are comfortable with technology-mediated interventions, may not yet have developed obesity-related illnesses, and contain a relatively high percentage of women compared to previous Veteran cohorts. Technology-mediated lifestyle interventions that include continuous, objective home monitoring of physical activity, automated internet mediated feedback, and e-coaching increase physical activity and improve weight loss in non-Veteran populations. When delivered on a large scale, such interventions represent low cost but effective alternatives to face-to-face lifestyle change interventions that can be implemented widely in the VA health care system. Thus, this project will test the feasibility and effectiveness of the prevention focused, internet-mediated healthy lifestyle physical activity program, Stay Strong w/coaching, tailored to the needs, preferences and demographics of OEF/OIF/OND Veterans. Specifically, Stay Strong w/coaching relies on use of a wearable device, the Fitbit Charge 2, and incorporates coaching support, tailored messages, and personalized physical activity goals. Stay Strong w/coaching will be compared to the use of the Fitbit Charge 2 with standard online support (Stay Strong).

ELIGIBILITY:
Inclusion Criteria:

1. OEF/OIF/OND Veteran
2. Can identify a VA Medical Center and VA Health Care Provider responsible for his/her care in the system
3. Interested in starting a physical activity program in the next 30 days
4. Access to a computer with an internet connection and a working USB port.
5. A smartphone running a compatible iOS or Android operating system.
6. Younger than Age 65

Exclusion Criteria:

1. Veteran self-reports that a health care provider has told the patient that it is currently unsafe to exercise in an unsupervised or unmonitored setting. (Can become eligible with written medical clearance).
2. History of eating disorders or a BMI < 20
3. Not competent to consent to a research study by self-reporting a legal guardian who makes medical decisions for the Veteran.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 465 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura J. Damschroder, MPH, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Buis LR, McCant FA, Gierisch JM, Bastian LA, Oddone EZ, Richardson CR, Kim HM, Evans R, Hooks G, Kadri R, White-Clark C, Damschroder LJ. Understanding the Effect of Adding Automated and Human Coaching to a Mobile Health Physical Activity App for Afghanistan and Iraq Veterans: Protocol for a Randomized Controlled Trial of the Stay Strong Intervention. JMIR Res Protoc. 2019 Jan 29;8(1):e12526. doi: 10.2196/12526. PMID 30694208
- [Derived] Olsen MK, Stechuchak KM, Hung A, Oddone EZ, Damschroder LJ, Edelman D, Maciejewski ML. A data-driven examination of which patients follow trial protocol. Contemp Clin Trials Commun. 2020 Aug 13;19:100631. doi: 10.1016/j.conctc.2020.100631. eCollection 2020 Sep. PMID 32913914
- [Derived] Damschroder LJ, Buis LR, McCant FA, Kim HM, Evans R, Oddone EZ, Bastian LA, Hooks G, Kadri R, White-Clark C, Richardson CR, Gierisch JM. Effect of Adding Telephone-Based Brief Coaching to an mHealth App (Stay Strong) for Promoting Physical Activity Among Veterans: Randomized Controlled Trial. J Med Internet Res. 2020 Aug 4;22(8):e19216. doi: 10.2196/19216. PMID 32687474
- [Derived] Buis LR, Dawood K, Kadri R, Dawood R, Richardson CR, Djuric Z, Sen A, Plegue M, Hutton D, Brody A, McNaughton CD, Brook RD, Levy P. Improving Blood Pressure Among African Americans With Hypertension Using a Mobile Health Approach (the MI-BP App): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2019 Jan 25;8(1):e12601. doi: 10.2196/12601. PMID 30681965

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Letters were mailed to potential participants. They used the information in the recruitment letter to accessed an online portal and respond to screening question. If eligible, they completed the consent documentation, baseline questionnaire, downloaded and registered the Stay Strong App. Recruitment period was from 10/1/2017 - 4/30/2018.
Pre-assignment Details: After consent and prior to randomization participants were to completed baseline survey, register app, and complete a baseline physical activity (PA) period for randomization. 56 participants were excluded due to failure to complete baseline survey or register app. 52 participants were excluded due to failure to provide baseline PA.
Period: Overall Study
Arm/Group | Stay Strong w/Coaching | Stay Strong
Started | 178 | 179
6month f/u Survey | 110 | 105
6month Physical Activity | 122 | 108
12month f/u Survey | 102 | 83
12month Physical Activity | 68 | 59
Completed | 102 | 83
Not Completed | 76 | 96
Not completed — Lost to Follow-up | 73 | 95
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Excluded | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stay Strong w/Coaching | Stay Strong | Total
Number analyzed (Participants) | 178 | 179 | 357
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (8.4) | 40.4 (9.0) | 39.8 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 43 | 90
  Male | 131 | 136 | 267
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic Black | 20 | 27 | 47
  Non-Hispanic White | 117 | 114 | 231
  Other | 41 | 38 | 79
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 178 | 179 | 357
Fitbit-Captured Active Minutes/Week, Median [Median (Inter-Quartile Range); unit: Active minutes/week] | 165 [75 to 328] | 190 [83 to 354] | 178 [80 to 346]
Fitbit-captured steps/day, mean [Mean (Standard Deviation); unit: Steps/day] | 7571 (3464) | 8163 (3978) | 7867 (3737)
Depression scale (PHQ-8), Median [Median (Inter-Quartile Range); unit: units on a scale] — Lower Scores Indicate a Better Outcome, Range: 0-24
  units on a scale | 7 [3 to 13] | 6 [3 to 11] | 6.5 [3 to 12]
Pain Intensity >=4 [Count of Participants; unit: Participants] | 80 | 75 | 155
PHQ-8 - Clinically Significant Depression [Count of Participants; unit: Participants] | 61 | 57 | 118

OUTCOME MEASURES:

1. Primary Outcome: Change in Physical Activity (PA) as Measured by the Study-provided Monitoring Device
Description: Physical activity is measured as Active Minutes by a wearable Fitbit Charge 2 device; daily activity is averaged over a one week period for which at least 5 days of valid data are available.
Time Frame: Change from Baseline in objectively monitored physical activity at one year after randomization
Population: Population decreases with time, at 12-month follow-up: SS+coaching 68; SS 58.
Measure: Least Squares Mean (95% Confidence Interval); unit: Active minutes/week
Arm/Group | Stay Strong w/Coaching | Stay Strong
Number analyzed (Participants) | 178 | 177
Active minutes/week | -67.1 [-141.5 to 7.35] | -69.0 [-148.1 to 10.18]
Statistical Analysis 1: Comparison: Stay Strong w/Coaching vs Stay Strong; Estimated marginal means/least squares means are derived from a linear mixed model/rmANOVA/rmANCOVA, adjusted for baseline AM goal, Type of Smart Phone, and Sex; Test type: Superiority; Slope = 1.88, 95% CI 2-sided [-119.0 to 122.7], Standard Error of Mean 46.2 — Generated through ANCOVA predicting Active Minutes as a function of arm and f/u time, adjusted for Sex, Baseline PA Goal (AM), and type of Smart Phone. Represents the contrast between SS+Coaching, 12 mos. - Baseline vs. SS alone, 12 mos. - Baseline

2. Secondary Outcome: Change in Weight as Measured From VA Medical Record
Description: Weights were extracted from VHA's Corporate Data Warehouse, vital signs package due to the high number of missing weights from the study provided blue tooth scale.
Time Frame: Change from Baseline in weight at one year after randomization
Population: Due to missing data from study provided scale, EHR weight was pulled for all patients, however, roughly half of the population lacked EHR weights within the time-frame of the study.
Measure: Least Squares Mean (95% Confidence Interval); unit: weight by pounds
Arm/Group | Stay Strong w/Coaching | Stay Strong
Number analyzed (Participants) | 32 | 33
weight by pounds | -0.121 [-7.25 to 7.01] | 4.902 [-1.65 to 11.45]
Statistical Analysis 1: Comparison: Stay Strong w/Coaching vs Stay Strong; The estimated marginal means/least squares means are derived from a linear mixed model/rmANOVA/rmANCOVA; Test type: Superiority; Slope = -5.02, 95% CI 2-sided [-15.85 to 5.81], Standard Error of Mean 56.7 — Generated through ANCOVA predicting Weight as a function of the interaction of arm and follow-up time. Estimate represents the contrast between SS+Coaching, 12 mos. - Baseline vs. SS alone, 12 mos. - Baseline

3. Secondary Outcome: Change in Depression Score as Assessed by the Personal Health Questionnaire Depression Scale (PHQ-8)
Description: The Personal Health Questionnaire Depression Scale (PHQ) will be administered via online survey. Personal Health Questionnaire (8 item version),Reporting Scores on a Scale Lower Scores Indicate a Better Outcome, Range: 0-24
Time Frame: Change from Baseline Depression score at one year after randomization
Population: Population decreases with time, at 12-month follow-up: SS+coaching 96; SS 81.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Stay Strong w/Coaching | Stay Strong
Number analyzed (Participants) | 170 | 168
score on a scale | -0.410 [-1.510 to 0.690] | 0.752 [-0.442 to 1.946]
Statistical Analysis 1: Comparison: Stay Strong w/Coaching vs Stay Strong; The estimated marginal means/least squares means are derived from a linear mixed model/rmANOVA/rmANCOVA; Test type: Superiority; Slope = -1.162, 95% CI 2-sided [-2.969 to 0.646], Standard Error of Mean 0.690 — Generated through ANCOVA predicting PHQ-8 Score as a function of the interaction of arm and follow-up time. Estimate represents the contrast between SS+Coaching, 12 mos. - Baseline vs. SS alone, 12 mos. - Baseline

4. Secondary Outcome: Change in Pain Measures as Assessed by the VA Pain Intensity
Description: Pain intensity will be elicited via online survey. Neuropathic Pain in Past Week Reporting Scores on a Scale, Lower Scores Indicate a Better Outcome, Range: 0-10
Time Frame: Change from Baseline in Pain measures at one year after randomization
Population: Population decreases with time, at 12-month follow-up: SS+coaching 101; SS 84.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Stay Strong w/Coaching | Stay Strong
Number analyzed (Participants) | 178 | 179
units on a scale | 0.212 [-0.215 to 0.639] | 0.557 [0.097 to 1.018]
Statistical Analysis 1: Comparison: Stay Strong w/Coaching vs Stay Strong; The estimated marginal means/least squares means are derived from a linear mixed model/rmANOVA/rmANCOVA; Test type: Superiority; Slope = -0.345, 95% CI 2-sided [-1.044 to 0.353], Standard Error of Mean 0.267 — Estimate generated through ANCOVA predicting "Pain In Past Week" as a function of the interaction of arm and follow-up time. Estimate represents the contrast between SS+Coaching, 12 mos. - Baseline vs. SS alone, 12 mos. - Baseline

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 1 year.
Description: Adverse event information was collected from participants if they reported events at quarterly status update. Adverse event information was also collected from patients through contact with coach interventionist or if patient reported during 6 or 12 month reminder calls for outcome survey. Adverse events were monitored/assessed without regard to the specific adverse event terms.
Arm/Group | Stay Strong w/Coaching | Stay Strong
All-Cause Mortality (participants affected / at risk) | 0/178 | 0/179
Serious Adverse Events (participants affected / at risk) | 0/178 | 0/179
Other Adverse Events (participants affected / at risk) | 3/178 | 1/179
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stay Strong w/Coaching (N=178) | Stay Strong (N=179)
Important Medical Event (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Important Medical Event (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Protocol Deviation (Investigations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Issue with device connectivity leading to missing data. PA is focused on proprietary measure of Active Minutes and any potential changes to how it is calculated by Fitbit are out of our control. Pain and Depression are self-reported measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-18): https://cdn.clinicaltrials.gov/large-docs/93/NCT02360293/Prot_SAP_000.pdf